CLINICAL TRIAL: NCT00320333
Title: Comparison of Pulmonary Rehabilitation of Patients With Chronic Obstructive Pulmonary Disease in Primary and Secondary Health Care
Brief Title: COPD Rehabilitation in Primary and Secondary Health Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Other Study IDs: 2004-53-1071
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; rehabilitation; health services research
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Procedure: pulmonary rehabilitation programme

SUMMARY:
Pulmonary rehabilitation of COPD patients are implemented in a non-randomized manner in two settings: primary and secondary health care. The effect on quality of life and hospitalizations will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* COPD patients

Exclusion Criteria:

* severe concomitant chronic disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2004-12; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Vest, MD, Principal Investigator — Glostrup University Hospital, Copenhagen; Allan Linneberg, MD, PhD, Study Chair — GloustrupUH
Locations (2):
- Denmark (2):
  - Omsorgscentret Kildegården, Gladsaxe, Gladsaxe
  - Department of Internal Medicin, Glostrup University Hospital, Copenhagen, Glostrup